CLINICAL TRIAL: NCT07399483
Title: Evaluation of the Biomechanical Response of Orthodontic Tooth Movement to Clear Aligner vs Fixed Orthodontic Appliance: A Randomized Clinical Trial
Brief Title: Evaluation of the Biomechanical Response of Orthodontic Tooth Movement to Clear Aligner vs Fixed Orthodontic Appliance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamad Alamin, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.25.08.67
Record Dates: First submitted 2025-12-24; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Orthodontic Tooth Movement; Tooth Movement
Keywords: Gingival crevicular fluid (GCF) Interleukin-1β (IL-1β) Prostaglandin E2 (PGE2) Cytokines Tooth mobility 3D digital superimposition; gingival cervical fluid , tooth mobility , Interleukin-1β (IL-1β) Prostaglandin E2; Gingival crevicular fluid (GCF) , Interleukin-1β (IL-1β) ,Prostaglandin E2 (PGE2), mobility test
MeSH Terms: conditions — Tooth Mobility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixed orthodontic appliance (Experimental): counting of Interleukin-1β and Prostaglandin E2 in gingival crevicular fluid, evaluation of the amount of tooth movement using intraoral scan and superimposition, tooth mobility using periotest devise and pain evaluation during orthodontic treatment
  Interventions: Diagnostic Test: diagnostic Test: Collection of GCF: from the gingival sulcus using paper point ,Tooth Mobility via Periotest ,3D Digital Model Superimposition using Intraoral Scanning
- clear aligner appliance (Experimental): counting of Interleukin-1β and Prostaglandin E2 in gingival crevicular fluid, evaluation of the amount of tooth movement using intraoral scan and superimposition, tooth mobility using periotest devise and pain evaluation during orthodontic treatment
  Interventions: Diagnostic Test: diagnostic Test: Collection of GCF: from the gingival sulcus using paper point ,Tooth Mobility via Periotest ,3D Digital Model Superimposition using Intraoral Scanning

INTERVENTIONS:
Diagnostic Test: diagnostic Test: Collection of GCF: from the gingival sulcus using paper point ,Tooth Mobility via Periotest ,3D Digital Model Superimposition using Intraoral Scanning — Diagnostic Tests Used in this Study
  1. Gingival Crevicular Fluid (GCF) Biomarker Analysis
     • Collection of GCF: GCF is collected from the gingival sulcus using absorbent paper points to obtain
  2. Tooth Mobility Measurement
     • Periotest Analysis: A mechanical diagnostic tool (Periotest device) that measures the damping characteristics of the periodontium by recording the reaction to a controlled tapping force is used
  3. 3D Digital Model Superimposition using intraoral scan device

SUMMARY:
Abstract

Background: Orthodontic tooth movement (OTM) is mediated by biologic responses of the periodontal ligament (PDL) and alveolar bone to applied mechanical forces, involving release of inflammatory mediators such as interleukin-1β (IL-1β) and prostaglandin E2 (PGE2) that promote osteoclast activation and bone remodeling. Intraoral biomarkers in gingival crevicular fluid (GCF) reflect these tissue changes and can be used to monitor inflammatory and metabolic responses during treatment. Digital technologies, including intraoral scanning and 3D superimposition, allow precise quantification of tooth movement over time.

Objective: This prospective, randomized comparative clinical study aims to compare the biological and mechanical responses of orthodontic tooth movement in patients treated with clear aligners versus conventional fixed appliances.

Methods: Twenty adult patients (aged 18-25 years) with mild dental crowding will be randomly assigned to either a fixed appliance group (n=10) or a clear aligner group (n=10). Baseline and follow-up GCF samples will be collected to quantify IL-1β and PGE2 using enzyme-linked immunosorbent assay (ELISA). Tooth mobility will be assessed using Periotest analysis, and 3D digital models obtained from intraoral scans will be superimposed to measure the amount of tooth movement over time. Secondary outcomes include clinical measures of mobility and patient-reported pain.

Expected Outcomes: It is anticipated that both treatment modalities will induce measurable increases in inflammatory biomarkers and tooth movement; however, differences in the magnitude and temporal patterns of IL-1β, PGE2, tooth mobility, and 3D-quantified displacement are expected due to the continuous forces of fixed appliances versus intermittent forces of aligners. Previous studies have shown that GCF cytokine levels rise with orthodontic force application in both aligner and fixed appliance treatments, with some variations between groups.

Conclusion: This study will provide new clinical evidence comparing biological mediator profiles and mechanical outcomes between clear aligners and fixed orthodontic appliances, improving understanding of tissue responses and informing clinical decision-making in contemporary orthodontic practice

DETAILED DESCRIPTION:
1. Introduction

   Orthodontic tooth movement (OTM) is a biologically mediated process that occurs as a response to mechanical forces applied to teeth. These forces should ideally be continuous and controlled, as they initiate cellular and molecular changes within the periodontal ligament (PDL) and surrounding alveolar bone. Mechanical loading results in vascular alterations within the PDL, followed by the release of inflammatory mediators that regulate bone modeling and remodeling. This cascade ultimately leads to osteoclastic bone resorption on the pressure side and osteoblastic bone formation on the tension side.

   Gingival crevicular fluid (GCF) is a serum transudate or inflammatory exudate originating from the gingival sulcus and was first described by Alfano. It serves as a valuable, non-invasive medium for monitoring biochemical changes occurring in the periodontium during orthodontic treatment. GCF contains a variety of biologically active molecules, including proteins, cytokines, bacterial antigens, enzymes, electrolytes, and small organic compounds derived from both host tissues and oral microorganisms.

   Application of orthodontic forces, particularly in the presence of plaque accumulation, induces a localized inflammatory response in periodontal tissues. This response is characterized by the activation and release of inflammatory cytokines such as matrix metalloproteinases (MMPs), interleukins (ILs), and tumor necrosis factor-alpha (TNF-α). Among these, Interleukin-1 (IL-1), particularly IL-1β, plays a central role in immune regulation and acute-phase inflammatory responses. During orthodontic tooth movement, IL-1β levels are significantly elevated in human gingival fibroblasts and GCF, reflecting increased osteoclastic activity.

   Prostaglandin E2 (PGE2) is another key inflammatory mediator involved in orthodontic tooth movement. Elevated levels of IL-1β and PGE2 are typically observed during the early phase of orthodontic treatment. IL-1β promotes osteoclast differentiation and activation, while PGE2 acts synergistically to enhance bone resorption. Together, these mediators facilitate tooth movement and alveolar bone remodeling.

   Orthodontic tooth movement occurs in distinct phases, including an initial phase, a lag phase, and a secondary phase. In the secondary phase, direct bone resorption predominates following the removal of hyalinized tissue via undermining resorption. During this period, the PDL space becomes widened, leading to increased tooth mobility. Tooth mobility is a physiological phenomenon resulting from the viscoelastic properties of the PDL and the structural characteristics of the alveolar bone. It is widely recognized that tooth mobility increases during active orthodontic treatment and gradually returns to baseline levels during the retention phase.

   Assessment of tooth mobility is an important clinical parameter used to evaluate periodontal support and biomechanical responses throughout orthodontic treatment. Monitoring changes in mobility can aid in predicting treatment outcomes, identifying potential risks, and preventing post-treatment relapse. However, limited data are available regarding long-term changes in tooth mobility from the initiation of orthodontic treatment through the retention phase.

   Advancements in digital orthodontics, including intraoral scanners, CAD/CAM systems, and 3D printing, have revolutionized orthodontic diagnosis and treatment planning. Digital study models have largely replaced conventional plaster casts due to their accuracy, efficiency, reduced storage requirements, and enhanced patient comfort. Virtual models allow for precise measurement, simulation, and superimposition, facilitating quantitative assessment of tooth movement over time.

   Three-dimensional superimposition of serial digital models enables accurate evaluation of orthodontic tooth movement by registering models within a common coordinate system. This approach is critical in contemporary orthodontics for assessing treatment efficiency and appliance performance.

   Clear aligner therapy has gained popularity due to increasing esthetic demands and patient comfort. Aligners deliver intermittent orthodontic forces, which may influence the biological response of periodontal tissues differently from continuous forces applied by fixed appliances. Although aligners offer advantages such as improved oral hygiene and esthetics, evidence regarding their influence on bone metabolism and inflammatory mediator production remains limited.

   Therefore, this study aims to compare the biological and mechanical responses associated with orthodontic tooth movement using clear aligners versus fixed orthodontic appliances by evaluating inflammatory biomarkers (IL-1β and PGE2), tooth mobility, and the amount of tooth movement assessed through 3D digital superimposition.
2. Aim of the Study

   The aim of this study is to compare the biological and mechanical responses of orthodontic tooth movement between patients treated with clear aligners and those treated with fixed pre-adjusted edgewise appliances, through assessment of:

   Inflammatory mediators (IL-1β and PGE2) in gingival crevicular fluid

   Tooth mobility

   Amount of tooth movement using 3D digital superimposition
3. Patients and Methods Study Design

   This study is designed as a prospective, randomized comparative clinical trial to evaluate and compare the effects of fixed orthodontic appliances and clear aligners on biological and mechanical parameters of orthodontic tooth movement.

   Sample Size

   Sample size calculation was performed using G*Power software (version 3.1.9.7) with a study power of 90%, a type I error rate of 5%, and a one-tailed statistical test. Based on an effect size (f = 1.4034537) derived from the study by Muhammad Abdullah Kamran et al., and mean IL-1β values of 21.45 ± 1.88 for fixed appliances and 18.29 ± 2.57 for clear aligners, the minimum sample size required was 18 patients. To compensate for potential dropouts, the sample size was increased to 20 patients.

   Participants will be equally divided into two groups:

   Group I (Fixed appliance group): 10 patients

   Group II (Clear aligner group): 10 patients

   Randomization

   Participants will be randomly allocated into one of the two study groups using a computer-generated randomization sequence. Allocation concealment will be ensured, and the clinician responsible for outcome assessment will be blinded to group assignment.

   Ethical Considerations

   Written informed consent will be obtained from all participants prior to enrollment

   The study protocol will be approved by the Research Ethics Committee of Mansoura University

   The study will be conducted in accordance with ethical guidelines and regulations
4. Methodology Initial Digital Records

   Baseline intraoral scans will be obtained using a digital intraoral scanner (e.g., iTero or TRIOS) to record the initial position of teeth and serve as a reference for 3D superimposition.

   Clear Aligner Group

   Digital treatment planning will be performed

   Aligners will be fabricated using thermoforming techniques

   A clear thermoplastic sheet (e.g., Duran) will be heated and pressure- or vacuum-formed over a 3D-printed model

   Aligners will be trimmed, finished, polished, and delivered to the patient

   Fixed Appliance Group

   Pre-adjusted edgewise brackets will be bonded

   Initial alignment and leveling will be performed using a 0.012-inch nickel-titanium archwire
5. Statistical Analysis

   Data will be statistically analyzed using appropriate parametric or non-parametric tests depending on data distribution. Significance will be set at p ≤ 0.05.
6. Duration of the Study

The study duration is estimated to range from 8 months to 1 year.

8. Cost

The estimated total cost of the study is 120,000 Egyptian Pounds.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients aged 18-25 years.

  * Skeletal class I mild dental crowding per arch (≤ 4 mm).
  * Good oral hygiene and no active periodontal disease.
  * Normal vertical SN-GOGN angle 32+- 3.

Exclusion Criteria:

* • Patients with severe crowding or spacing (> 4 mm).

  * Presence of active dental caries or periodontal disease.
  * History of orthodontic treatment within the past two years.
  * Systemic conditions affecting tooth movement (e.g., diabetes, bone disorders).
  * Bimaxillary protrusion, sever proclination

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Interleukin-1β and Prostaglandin E2 | 4 week
  counting of Interleukin-1β and Prostaglandin E2 in gingival crevicular fluid

SECONDARY OUTCOMES:
amount of tooth movement | 4 weeks
  intraoral scan will be taken before and after movement, then superimposition will be done to measure the amount of tooth movement
tooth mobility | 4 weeks
  periotest devise will be used to measure the amount of tooth mobility
pain evaluation | 2 weeks
  pain evaluation will be done using visual analogue scale and health related quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Alamin Ahmed Elmansor, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, El Mansoura, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No